CLINICAL TRIAL: NCT07374289
Title: The Effectiveness of ECPR on the Scene and in Hospital for Out-of-hospital Cardi-ac Arrest (OHCA) in the Moravian-Silesian Region.
Brief Title: On Scene ECPR in Ostrava
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: Emergency Medical Services, Moravian-Silesian Region (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-KARIM-On-Scene-ECPR
Record Dates: First submitted 2026-01-09; First posted 2026-01-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Arrest (CA); Cardiogenic Shock
Keywords: extracorporeal membrane oxygenation; out-of-hospital cardiac arrest; cardiac arrest; cardiogenic shock
MeSH Terms: conditions — Heart Arrest; Shock, Cardiogenic; Out-of-Hospital Cardiac Arrest | interventions — Parturition

STUDY DESIGN:
Intervention Model Description: The study subjects will be enrolled in two parallel arms
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECPR on scene (Experimental): On-scene ECPR cannulation by mobile ECMO team according to protocol if the location of the arrest and circumstances appear to be suitable (distance from the ECMO centre, transport logistics, in an ambulance/at home, etc.)
  Interventions: Procedure: Prehospital ECMO cannulation on scene of cardiac arrest
- ECPR in hospital (Active Comparator): Hospital ECPR cannulation at Emergency Department by ECMO team accord-ing to protocol if a on scene ECPR call-out was not indicated.
  Interventions: Procedure: Transfer with ongoing mechanical chest compression to hospital followed by hospital ECMO cannulation

INTERVENTIONS:
Procedure: Prehospital ECMO cannulation on scene of cardiac arrest — ECPR (Extracorporeal Cardiopulmonary Resuscitation) is a critical, advanced resuscitation technique using Veno-arterial Extracorporeal Membrane Oxygenation for patients in cardiac arrest where conventional CPR fails, functioning as a bridge to restore circulation and oxygenation by pumping and oxygenating blood outside the body before returning it.
  Arms: ECPR on scene
Procedure: Transfer with ongoing mechanical chest compression to hospital followed by hospital ECMO cannulation — ECPR (Extracorporeal Cardiopulmonary Resuscitation) is a critical, advanced resuscitation technique using Veno-arterial Extracorporeal Membrane Oxygenation for patients in cardiac arrest where conventional CPR fails, functioning as a bridge to restore circulation and oxygenation by pumping and oxygenating blood outside the body before returning it.
  Arms: ECPR in hospital

SUMMARY:
On-scene extracorporeal pulmonary resuscitation (ECPR) for out-of-hospital cardiac arrest (OHCA) seems to speed up the start of extracorporeal membrane oxygenation (ECMO) and shorten low flow during cardiopulmonary resuscitation (CPR) in case of refractory cardiac arrest. The primary goal is to verify the benefit of on-scene ECPR in terms of shortening the collapse-to-ECMO interval. The secondary goal is to compare outcomes in the on-scene ECPR group with hospital cannulation.

DETAILED DESCRIPTION:
ECPR is a life-saving method for a selected group of patients who are refractory to standard resuscitation procedures. With the appropriate use of ECPR, it is possible to achieve a significant improvement in survival with good neurological outcomes even in patients who would otherwise die. The ECMO Centre Ostrava has been providing ECPR for OHCA since 2022 with cannulation in the hospital after prior transport from the scene under continuous resuscitation. A good neurological outcome is achieved in approximately 29% of patients, even though the collapse-ECMO interval is around 75 minutes. Shortening this interval, which is associated with improved outcomes, is possible by using a mobile team that per-forms cannulation directly on scene. Mobile ECPR will be carried out in cooperation with the Ostrava University Hospital and the Moravian-Silesian Region Emergency Medical Service. The primary objective is to verify the benefit of on-scene ECPR in terms of shortening the collapse-ECMO interval. The secondary objective is to compare the outcome in the on-scene ECPR group with hospital cannulation.

ELIGIBILITY:
Inclusion Criteria:

* Presumed cardiac aetiology of the cardiac arrest
* Witnessed collapse
* Bystander CPR
* Estimated age ≤ 70 years
* Body weight ≥15 Kg

Exclusion Criteria:

* Known terminal malignant disease
* Known terminal chronic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital survival | 30 days after the cardiac arrest
  Hospital survival will be assessed 30 days after the cardiac arrest
ICU stay | Through the ICU stay, on average 12 days
  The length of the Intensive Care Unit (ICU) stay will be assessed in days.
Neurologic outcomes | 30 days after the cardiac arrest
  Neurologic outcomes will be assessed in patients using the Cerebral Performance Category (CPC) score. The CPC score is a 1-to-5 scale assessing neurological outcome, most commonly after cardiac arrest, where 1 is best (normal brain function) and 5 is worst (brain death).

SECONDARY OUTCOMES:
Collapse to ECMO interval | One hour
  The interval from the collapse (cardiac arrest) to ECMO initiation will be measured in minutes.
Collapse to ECMO interval | From the collapse (cardiac arrest) to ECMO initiation
  The interval from the collapse (cardiac arrest) to ECMO initiation will be measured in minutes.
Long-term outcome - Survival | 6 months after the collapse
  The long-term survival of patients will be assessed 6 months after the collapse.
Long-term outcome - Quality of Life | 6 months after the collapse
  Long-term quality of life will be assessed 6 months after the collapse using standardised tools (questionnaires).

CONTACTS AND LOCATIONS:
Overall Officials: Filip Burša, MD, PhD, EDEC, Principal Investigator — University Hospital Ostrava
Locations (2):
- Czechia (2):
  - Emergency Medical Services, Moravian-Silesian Region, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon reasonable request.